CLINICAL TRIAL: NCT01985594
Title: STUDY ON EFFICACY OF UTROGESTAN AS TOCOLYSIS FOR PRETERM LABOR
Brief Title: Utrogestan Versus Nifedipine as Tocolysis for Preterm Labor: a Randomised Controlled Trial
Acronym: UTROGESTAN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: nor zila hassan malek (Other)
Responsible Party: Sponsor-Investigator, nor zila hassan malek, medical officer, National University of Malaysia
Organization: National University of Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FF-2013-407
Record Dates: First submitted 2013-11-04; First posted 2013-11-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Preterm Labor
Keywords: preterm labor
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Utrogestan; Nifedipine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Utrogestan (Active Comparator): oral tablet Utrogestan 400mg daily for 2 days
  Interventions: Drug: utrogestan
- Nifedipine (Placebo Comparator): tablet Nifedipine 20 mg stat then 20 mg after 30 minutes then another 20 mg after 30 minutes followed by 10 mg three times daily for 2 days
  Interventions: Drug: Nifedipine

INTERVENTIONS:
Drug: utrogestan — Oral Tablet Utrogestan 400 mg daily for 2 days
  Arms: Utrogestan
Drug: Nifedipine — Tablet Nifedipine 20 mg stat then 20 mg after 30 minutes if contraction persist and another 20mg after 30 minutes if contraction still persist followed by 10 mg three times daily for 2 days
  Arms: Nifedipine

SUMMARY:
RESEARCH HYPOTHESIS

-Incidence of preterm delivery is lower in women treated with oral micronized progesterone (Utrogestan) as acute tocolysis agent compare to Nifedipine group with fewer maternal side effect

ELIGIBILITY:
Inclusion Criteria:

• Singleton pregnancy women between 22 and 34 weeks of gestation who presented with threatened preterm labor.

Exclusion Criteria:

* Multiple pregnancies
* Women with Preterm Prelabour Rupture of Membrane
* Fetal death
* Women with bad obstetric history
* Women with history of cervical incompetence
* Contraindication to Nifedipine such as cardiovascular disease, hyperthyroidism, severe pre eclampsia or to Utrogestan
* Maternal or fetal indication for immediate delivery, such as fetal distress, bleeding placenta previa, abruption placenta
* Contraindication for tocolysis, for example severe pre eclampsia, intrauterine growth restriction, fetal anomaly, chorioamnionitis, significant antepartum haemorrhage
* Cervical dilatation of 3cm or more
* Patients with previous tocolytic treatment during this pregnancy
* Women who refuse to participate in this study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-07 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
latency period interval between time of tocolysis and delivery | 24 hours up to 7 days
  delivery less than 24 hours of tocolysis,delivery less than 48 hours of tocolysis, delivery less than 7 days of tocolysis

SECONDARY OUTCOMES:
Pregnancy outcomes | 34 weeks of gestational age
  delivery less than 34 weeks of gestation, delivery more than or at 34 weeks of gestation
Neonatal outcome | 24 hours
  Birth weight (kg),cord blood acidity, need for neonatal intensive care unit admission
Maternal side effect | 30 minutes up to 48 hours
  Palpitation,Headache, Nausea/Vomiting, Hypotension, Dyspnea, Jaundice, Pruritus

CONTACTS AND LOCATIONS:
Overall Officials: nor azlin mohamed ismail, Principal Investigator — National University of Malaysia
Locations (1):
- Obstetric and Gynaecology Department, National University of Malaysia Medical Centre, Cheras, Kuala Lumpur, Malaysia

REFERENCES:
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046